CLINICAL TRIAL: NCT07340788
Title: Amylin-Induced Migraine Attacks Without Aura: A Randomized Clinical Trial
Brief Title: Amylin-Induced Migraine Attacks Without Aura
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Håkan Ashina, Associate Professor, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-24025082
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Headache Disorders, Primary; Headache Disorders; Brain Diseases; Nervous System Diseases; Central Nervous System Diseases; Neurologic Manifestations; Signs and Symptoms; Pathological Conditions, Signs and Symptoms; Migraine Disorders; Headache; Pain; Peptide Hormones; Hormones; Hormones, Hormone Substitutes, and Hormone Antagonists; Peptides; Amino Acids, Peptides, and Proteins; Amylin; Pramlintide
Keywords: Migraine; Headache; Pain; Amylin
MeSH Terms: conditions — Headache Disorders, Primary; Headache Disorders; Brain Diseases; Nervous System Diseases; Central Nervous System Diseases; Neurologic Manifestations; Signs and Symptoms; Pathological Conditions, Signs and Symptoms; Migraine Disorders; Headache; Pain | interventions — Islet Amyloid Polypeptide

STUDY DESIGN:
Intervention Model Description: This single-center trial applies a randomized, double-blind, placebo-controlled, two-way crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amylin (Experimental): Pramlintide (Amylin) will be administered by intravenous infusion.
  Interventions: Drug: Amylin
- Placebo (Placebo Comparator): Placebo (isotonic saline) will be administered by intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amylin — The participants will receive continuous intravenous infusion of 20 mL (6 μg/min) of pramlintide (amylin) over 20 minutes.
  Arms: Amylin
Drug: Placebo — The participants will receive continuous intravenous infusion of 20 mL of placebo (isotonic saline) over 20 minutes.
  Arms: Placebo

SUMMARY:
Pramlintide is a peptide analogue of human amylin which is a vasoactive signaling molecule involved in the pathogenesis of migraine. This study investigates whether pramlintide induces migraine attacks without aura in people with migraine without aura.

DETAILED DESCRIPTION:
Amylin is a vasoactive substance that acts on vascular smooth muscle and can cause vasodilation. It is naturally present in the trigeminovascular system, an important structure involved in headache development. Recent studies indicate that intravenous infusion of pramlintide, an amylin analogue, can trigger migraine attacks in people with migraine. This study aims to determine whether intravenous pramlintide can induce migraine attacks without aura in individuals who experience migraine without aura. To test this, the investigators will conduct a randomized, double-blind, placebo-controlled, two-way crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age upon entry into screening
* A body weight of 50 to 100 kg
* History of migraine without aura for ≥12 months and in accordance with ICHD-3
* Between 1-5 monthly migraine days without aura on average across the 3 months prior to screening
* Provision of informed consent prior to initiation of any study-specific activities/procedures

Exclusion Criteria:

* Any history of a primary or secondary headache disorder other than migraine without aura and infrequent episodic tension-type headache
* Any history of moderate to severe traumatic brain injury
* Any history of cardiovascular disease, including cerebrovascular diseases
* Any history of pulmonary disease
* Any other clinically significant disorders, conditions, or diseases that might impact the safety of the subject or interfere with the study's evaluation, procedures, or completion, aside from those mentioned above. This includes any relevant medical history or evidence that, in the opinion of the site investigator, might pose a risk to the subject or impact the validity of the study results
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior
* Female subjects of childbearing potential with a positive pregnancy test during any study visit
* Cardiovascular disease of any kind, including cerebrovascular diseases
* Hypertension (systolic blood pressure of ≥150 mmHg and/or diastolic blood pressure of ≥100 mmHg) prior to the start of infusion on the experimental day
* Hypotension (systolic blood pressure of ≤90 mmHg and/or diastolic blood pressure of ≤50 mmHg)
* Abnormalities on the electrocardiogram that, in the opinion of the site investigator, might pose a risk to the subject or impact the validity of the study results
* Daily use of any medication other than contraceptives
* Intake of any medication other than contraceptives within 48 hours of infusion start
* Intake of caffeine, nicotine, and alcohol within 12 hours of infusion start
* Headache of any intensity within 48 hours of infusion start
* Migraine attack within 48 hours of infusion start
* Aura within 48 hours of infusion start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of migraine attacks without aura | 12 hours
  The difference in the incidence of migraine attacks without aura between pramlintide and placebo during the 12-hour observational period after infusion start.

SECONDARY OUTCOMES:
Headache intensity scores | 12 hours
  The secondary outcome is the difference in the area under the curve (AUC) for median headache intensity scores between pramlintide and placebo during the 12-hour observational period after infusion start.

OTHER OUTCOMES:
Superficial temporal artery dilation | 2 hours
  The difference in AUC for relative superficial temporal artery (STA) dilation between pramlintide and placebo from the start of infusion to 2 hours after the infusion.
Middle cerebral artery blood flow velocity | 2 hours
  The difference in AUC for change in middle cerebral artery (MCA) mean blood flow velocity between pramlintide and placebo from the start of infusion to 2 hours after the infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: Anonymized data not published within this article will be made available on reasonable request from any qualified investigator.

REFERENCES:
- [Background] Asmar M, Bache M, Knop FK, Madsbad S, Holst JJ. Do the actions of glucagon-like peptide-1 on gastric emptying, appetite, and food intake involve release of amylin in humans? J Clin Endocrinol Metab. 2010 May;95(5):2367-75. doi: 10.1210/jc.2009-2133. Epub 2010 Mar 1. PMID 20194711
- [Background] Hay DL, Chen S, Lutz TA, Parkes DG, Roth JD. Amylin: Pharmacology, Physiology, and Clinical Potential. Pharmacol Rev. 2015 Jul;67(3):564-600. doi: 10.1124/pr.115.010629. PMID 26071095
- [Background] Ghanizada H, Al-Karagholi MA, Walker CS, Arngrim N, Rees T, Petersen J, Siow A, Morch-Rasmussen M, Tan S, O'Carroll SJ, Harris P, Skovgaard LT, Jorgensen NR, Brimble M, Waite JS, Rea BJ, Sowers LP, Russo AF, Hay DL, Ashina M. Amylin Analog Pramlintide Induces Migraine-like Attacks in Patients. Ann Neurol. 2021 Jun;89(6):1157-1171. doi: 10.1002/ana.26072. Epub 2021 Apr 8. PMID 33772845
- [Background] Hansen JM, Hauge AW, Olesen J, Ashina M. Calcitonin gene-related peptide triggers migraine-like attacks in patients with migraine with aura. Cephalalgia. 2010 Oct;30(10):1179-86. doi: 10.1177/0333102410368444. Epub 2010 May 12. PMID 20855363
- [Background] Ashina M, Hansen JM, Do TP, Melo-Carrillo A, Burstein R, Moskowitz MA. Migraine and the trigeminovascular system-40 years and counting. Lancet Neurol. 2019 Aug;18(8):795-804. doi: 10.1016/S1474-4422(19)30185-1. Epub 2019 May 31. PMID 31160203
- [Background] Ashina M, Terwindt GM, Al-Karagholi MA, de Boer I, Lee MJ, Hay DL, Schulte LH, Hadjikhani N, Sinclair AJ, Ashina H, Schwedt TJ, Goadsby PJ. Migraine: disease characterisation, biomarkers, and precision medicine. Lancet. 2021 Apr 17;397(10283):1496-1504. doi: 10.1016/S0140-6736(20)32162-0. Epub 2021 Mar 25. PMID 33773610
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Ashina M. Migraine. N Engl J Med. 2020 Nov 5;383(19):1866-1876. doi: 10.1056/NEJMra1915327. No abstract available. PMID 33211930
- See also: Related Info — https://www.regionh.dk/til-fagfolk/forskning-og-innovation/de-regionale-videnskabsetiske-komiteer/sider/default.aspx